CLINICAL TRIAL: NCT04833504
Title: Clinical Follow-up Study of CD19 CAR-T Expressing IL7 and CCL19 for Relapsed or Refractory B Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: I20200011057
Record Dates: First submitted 2020-12-14; First posted 2021-04-06 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2021-01

CONDITIONS: Diffuse Large B-cell Lymphoma; Mantle Cell Lymphoma; Transformed Follicular Lymphoma; Primary Mediastinal Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: CD19 CAR-T Expressing IL7 and CCL19 — A fourth generation CD19 targeting CAR-T expressing IL7 and CCL19

SUMMARY:
This study is designed to monitor all patients exposed to CD19 CAR-T expressing IL7 and CCL19 for 5 years following infusion, to assess their long-term efficacy, including the CAR-vector persistence, the normal immunity rebuilding and the risk of delayed adverse events (AEs).

DETAILED DESCRIPTION:
Patients are enrolled following completion from the early clinical study of CD19-7X19 CAR-T treatment ( NCT03258047) and will be followed for 5 years post treatment from the last treatment. They will be monitored for safety and efficacy with the primary treatment protocols for the protocol defined duration. This long-term following up study allow an interim analysis to evaluate the outcomes of the study when it arrives in 2 years Collection of such long term effects of CAR-T cell therapy will help to further define the risk-benefit profile of CAR-T Therapies.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have received the CD19-IL7/CCL19 CAR-T therapy in the earlier enrolled clinical trail and met including and excluding criteria criteria (NCT0325847) Patients who have provided informed consent for the long term follow up study prior to their study participation .

Exclusion Criteria:

* There are no specific exclusion criteria for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 39 patients meet including and excluding criteria criteria
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2018-09-22 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of CD19-IL7/CCL19 CAR-T | 5 years
  Evaluate the efficacy of CD19-IL7/CCL19 CAR-T including duration of response, progression-free survival, overall surviva and objective response rate (CR + PR) .

SECONDARY OUTCOMES:
Evaluate the persistence of CAR-T cells | 5 years
  Levels and persistence of CAR+ T cells in serum samples
Evaluate the incidence of adverse events | 5 years
  The incidence of CRS and CRES; Levels and persistence of cytokines in serum samples;Proportion of patients who relapse or progress among patients who had not relapsed or progressed at study entry/re-entry;Incidence of death ;B- and T- lymphocyte count;

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Qian, Doctor, Study Chair — Zhejiang University
Locations (1):
- Hui Liu, Hangzhou, State..., China